CLINICAL TRIAL: NCT05750147
Title: Genetics, Imaging and Artificial Intelligence for Precision Care in Cardiomyopathy
Brief Title: The SMARTER Cardiomyopathy Study
Acronym: SMARTER-CM
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 22IC7783
Record Dates: First submitted 2023-01-23; First posted 2023-03-01 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Cardiomyopathies; Hypertrophic Cardiomyopathy; Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies; Cardiomyopathy, Hypertrophic; Cardiomyopathy, Dilated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Blood- plasma and serum
  2. Saliva
  3. Collection of additional tissue samples (myocardial, skeletal, skin) or excess diagnostic materials from planned clinical procedures (where applicable)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiomyopathies: Approximately 1000 participants recruited prospectively from participating sites with a diagnosis of cardiomyopathy
  Participants will provide biosamples and allow access to medical scans and records for health data collection
  Interventions: Other: Blood Sample Collection

INTERVENTIONS:
Other: Blood Sample Collection — Blood for DNA and biomarker analysis

SUMMARY:
Cardiomyopathies are diseases of the heart muscle. Known genetic factors may account for some cardiomyopathy cases but there is still much to understand about the genetic and environmental causes and how the disease progresses.

Finding new ways to diagnose and treat cardiomyopathies could improve the health and well-being of patients with these conditions.

This study will collect data from individuals with cardiomyopathy or related heart muscle disease, or with a possible genetic predisposition to cardiomyopathy, and follow them over time to observe the progress of their heart and health. This study will collect DNA, blood samples, and detailed clinical & lifestyle information at the start of the study, and data collected during routine healthcare visits over time.

* learn what causes cardiomyopathy, and therefore how to treat it
* understand why cardiomyopathy progresses differently in different people, to improve the ability to recognise who will benefit from different treatments at different times

The investigators will collaborate with other centres internationally to collect a large of group of participants with similar cardiomyopathies, providing power to identify new pathways that cause disease and ways of predicting which participants are at risk of having more severe disease.

ELIGIBILITY:
Inclusion Criteria:

Adults with the capacity to consent Children with parental/guardian consent Male and Female

Meeting the following criteria:

1. Patients with a confirmed diagnosis of cardiomyopathy or related condition
2. Patients with a family member with cardiomyopathy, or a related condition
3. Patients with a genetic variant that may predispose to cardiomyopathy, or a related condition

Exclusion Criteria:

Patients without the capacity to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with a diagnosis of cardiomyopathy, or a family member of cardiomyopathy or a genetic predisposition to cardiomyopathy of any age and any sex.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of genetic variants | 5 years
  Rare and common genetic variants in people with cardiomyopathy
The incidence of major adverse cardiovascular events over 5 years | 5 years
  The incidence of major adverse cardiovascular events over 5 years, defined as:-
  1. Cardiovascular death
  2. Major arrhythmic events (ventricular fibrillation, unstable sustained ventricular tachycardia, appropriate implantable cardioverter-defibrillator delivered shock, and aborted sudden cardiac death)
  3. Major heart failure events (heart transplantation, left ventricular assist device implantation, unplanned heart failure hospitalisation)

CONTACTS AND LOCATIONS:
Overall Officials: James Ware, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Guys & St Thomas' NHS Foundation Trust, London
  - Kings College Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with collaborating researchers in a pseudonymised fashion (removing names, addresses, identifying numbers, DOB etc)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: During study duration (Aug 2027)
Access Criteria: Provided through secure data transfer mechanisms approved by Imperial College London, following full GDPR (data protection) assessments and collaborating agreements.